CLINICAL TRIAL: NCT03628807
Title: Non-invasive Evaluation of Prognostic Parameters for Patients With Transjugular Intrahepatic Portosystemic Shunt (TIPS) Using a Structured Follow up Protocol
Brief Title: Non-invasive Evaluation Program for TIPS and Follow Up Network
Acronym: NEPTUN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Jonel Trebicka, Professor, University Hospital, Bonn
Other Study IDs: NEPTUN
Record Dates: First submitted 2018-07-11; First posted 2018-08-14 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Portal Hypertension
Keywords: transjugular intrahepatic portosystemic shunt (TIPS); non-invasive assessments; Transthoracic echocardiography (TTE) with Speckle-tracking; Computer tomography scan (CT-scan); Magnetic resonance imaging (MRI); circulating biomarkers; Electroencephalography (EEG)
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — serum, plasma, stool, DNA, PBMC, Buffi coat
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective 1: Retrospective Bare Metal Stent Cohort that received TIPS from 01/01/1996 to 12/31/2003.
- Retrospective 2: Retrospective Covered Stent Cohort that received TIPS from 01/01/2004 to 12/31/2012.
- Prospective: Prospective cohort that received TIPS from 01/01/2013 onwards

SUMMARY:
Evaluation of non-invasive prognostic parameters in patients receiving transjugular intrahepatic portosystemic shunt (TIPS) for complications of portal hypertension. Patients are cared according to the local standardized follow up program. Clinical and laboratory data from standard patient care are evaluated for potential prognostic value.

DETAILED DESCRIPTION:
NEPTUN consists of liver cirrhosis receiving transjugular intrahepatic portosystemic shunt (TIPS) at the Department of Internal Medicine I, University of Bonn, Germany and receiving a structured routine evaluation and follow up program. The diagnosis of cirrhosis was based on clinical, hemodynamic and biochemical parameters, and ultrasound and/or biopsy criteria.

ELIGIBILITY:
Inclusion Criteria:

* Insertion of TIPS according to guidelines

Exclusion Criteria:

* Contraindication for TIPS

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving TIPS according to guidelines
Sampling Method: Non-Probability Sample
Enrollment: 747 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Survival | up to 10 years
  death, liver transplantation

SECONDARY OUTCOMES:
Ascites | up to 10 years
  Evaluation of amount of ascites according to the Child-Score
Hepatic Encephalopathy | up to 10 years
  Evaluation of the grade according to the West Haven Criteria
Variceal Bleeding | up to 10 years
  Assessment of presence of variceal bleeding
Liver Failure | up to 10 years
  defined as Bilirubin level ≥ 12mg/dl
Acute-on-Chronic-Liver Failure (ACLF) | up to 10 years
  Presence of ACLF according to the EASL-Chronic liver Failure Consortium (CLIF)-criteria
Organ Failures | up to 10 years
  Assessment of Organ failures according to the CLIF-SOFA
  according to CLIF-Sequential Organ Failure Assessment (SOFA) Score

CONTACTS AND LOCATIONS:
Overall Officials: Michael Praktiknjo, MD, Principal Investigator — University of Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany

REFERENCES:
- [Derived] Meyer C, Kimmann M, Bohm K, Nowak S, Perez AMP, Meier JA, Reinartz Groba SN, Godiker J, Uschner FE, Sanoubara F, Chang J, Trebicka J, Sprinkart AM, Praktiknjo M. Three-Dimensional Transjugular Intrahepatic Portosystemic Shunt Geometry Predicts Shunt Dysfunction. Aliment Pharmacol Ther. 2025 Jun;61(11):1805-1814. doi: 10.1111/apt.70133. Epub 2025 Apr 9. PMID 40202365
- [Derived] Queck A, Schwierz L, Gu W, Ferstl PG, Jansen C, Uschner FE, Praktiknjo M, Chang J, Brol MJ, Schepis F, Merli M, Strassburg CP, Lehmann J, Meyer C, Trebicka J. Targeted decrease of portal hepatic pressure gradient improves ascites control after TIPS. Hepatology. 2023 Feb 1;77(2):466-475. doi: 10.1002/hep.32676. Epub 2022 Aug 12. PMID 35869810
- [Derived] Praktiknjo M, Abu-Omar J, Chang J, Thomas D, Jansen C, Kupczyk P, Schepis F, Garcia-Pagan JC, Merli M, Meyer C, Strassburg CP, Pieper CC, Trebicka J. Controlled underdilation using novel VIATORR(R) controlled expansion stents improves survival after transjugular intrahepatic portosystemic shunt implantation. JHEP Rep. 2021 Mar 3;3(3):100264. doi: 10.1016/j.jhepr.2021.100264. eCollection 2021 Jun. PMID 34013182
- [Derived] Torner M, Mangal A, Scharnagl H, Jansen C, Praktiknjo M, Queck A, Gu W, Schierwagen R, Lehmann J, Uschner FE, Graf C, Strassburg CP, Fernandez J, Stojakovic T, Woitas R, Trebicka J. Sex specificity of kidney markers to assess prognosis in cirrhotic patients with TIPS. Liver Int. 2020 Jan;40(1):186-193. doi: 10.1111/liv.14230. Epub 2019 Sep 10. PMID 31448496
- [Derived] Lehmann J, Praktiknjo M, Nielsen MJ, Schierwagen R, Meyer C, Thomas D, Violi F, Strassburg CP, Bendtsen F, Moller S, Krag A, Karsdal MA, Leeming DJ, Trebicka J. Collagen type IV remodelling gender-specifically predicts mortality in decompensated cirrhosis. Liver Int. 2019 May;39(5):885-893. doi: 10.1111/liv.14070. Epub 2019 Mar 7. PMID 30739387